CLINICAL TRIAL: NCT05032066
Title: A Phase 2b Randomized, Double-blind, Placebo-controlled, Repeat-dose, Multicenter Trial to Evaluate the Efficacy, Safety and Tolerability of HZN-825 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Multicenter Trial to Evaluate the Efficacy, Safety and Tolerability of HZN-825 in Subjects With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated due to not meeting primary or key secondary endpoints.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HZNP-HZN-825-303; 2023-509784-24-00 (EU CTIS Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- HZN-825 300 mg once daily (QD) (Experimental): Two 150 mg oral tablets given in the morning with a meal and two matching placebo tablets given in the evening with a meal; total daily dose 300 mg HZN-825.
  Interventions: Drug: HZN-825
- HZN-825-300 mg twice daily (BID) (Experimental): Two 150 mg oral tablets given in the morning with a meal and two 150 mg oral tablets given in the evening with a meal; total daily dose 600 mg HZN-825.
  Interventions: Drug: HZN-825
- Placebo BID (Placebo Comparator): Matching placebo tablets (2) given in the morning with a meal and matching placebo tablets (2) given in the evening with a meal; total dose 4 placebo tablets.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HZN-825 — Core Phase: Participants will receive HZN-825 300 mg QD, HZN-825 300 mg BID or matching placebo orally in the morning and evening with a meal for 52 weeks according to randomization schema.
  Extension Phase: Participants will receive open-label HZN-825 150 mg orally in the morning and evening with a meal for 52 weeks.
  Arms: HZN-825 300 mg once daily (QD); HZN-825-300 mg twice daily (BID)
Drug: Placebo — Core Phase: Participants will receive HZN-825 300 mg QD, HZN-825 300 mg BID or matching placebo orally in the morning and evening with a meal for 52 weeks according to randomization schema.
  Extension Phase: Participants who received matching placebo in the Core Phase will receive open-label HZN-825 150 mg orally in the morning and evening with a meal for 52 weeks.
  Arms: Placebo BID

SUMMARY:
HZNP-HZN-825-303 (HARBOR) comprises of 2 parts. Part 1 (Core Phase) is a randomized, double-blind, placebo-controlled, repeat-dose, multicenter trial to evaluate the efficacy, safety and tolerability of HZN-825 in participants with Idiopathic Pulmonary Fibrosis (IPF).

Part 2 (Extension Phase) is an optional, open-label, repeat-dose, multicenter extension of the Core Phase. The trial will include up to an 8-week Screening Period and a 52-week Double-blind Treatment Period in the Core Phase and 52 weeks of open-label HZN-825 treatment in the Extension Phase.

During the Core Phase, participants will be screened within 8 weeks prior to the baseline (Day 1) Visit. Approximately 135 participants who meet the trial eligibility criteria will be randomly assigned in a 1:1:1 ratio on Day 1 to receive HZN-825 300 mg QD, HZN-825 300 mg BID or matching placebo orally for 52 weeks using the following 2 stratification factors:

1. Concomitant use of approved IPF therapy (i.e., nintedanib or pirfenidone): yes or no
2. Forced vital capacity (FVC) % predicted at Baseline: ≥70% or <70%

Participants who complete the 52-week Double blind Treatment Period of the Core Phase of the trial will be invited to extend their participation in the 52-week Extension Phase of the trial.

DETAILED DESCRIPTION:
Part 1 (Core Phase) The overall objective of the Core Phase is to investigate the efficacy, safety and tolerability of 2 dose regimens of HZN-825, a selective antagonist of lysophosphatidic acid receptor-1 (LPAR1), administered orally once daily (QD) or twice daily (BID) for 52 weeks in the treatment of participants with IPF.

Part 2 (Extension Phase) The overall objective of the Extension Phase is to investigate the long-term efficacy, safety and tolerability of HZN-825, a selective antagonist of LPAR1, administered at a dose of 300 mg BID orally to participants with IPF in a 52-week open-label extension (OLE) following completion of the Core Phase of the trial. The dose for the Extension Phase may be modified based on the results of the Core Phase.

Two types of Baseline are defined for the Extension Phase:

* OLE Baseline, defined as the latest measurement prior to the first dose of HZN-825 in the Extension Phase
* HZN-825 Baseline, defined as the latest measurement prior to the first dose of HZN-825 in either the Core Phase or the Extension Phase. For subjects who received placebo in the Core Phase, OLE Baseline will be the same as HZN-825 Baseline.

Acquired from Horizon in 2024

ELIGIBILITY:
Key Inclusion Criteria in Core Phase:

1. Male or female ≥18 years of age at Screening.
2. Current diagnosis of IPF, as defined by American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Society (ALAT) guidelines and determined by central review; the date of initial diagnosis of IPF should be ≤7 years prior to Screening.
3. No recent changes or planned changes to the dose or regimen for IPF therapy, defined as:

   * Receiving a stable dose of IPF-approved therapy (i.e., nintedanib or pirfenidone) for a minimum of 3 months prior to Day 1 with no plans to change the background regimen during trial participation, or
   * Not currently receiving background IPF-approved therapy at Screening (either naïve to IPF-approved therapy or previously discontinued any IPF-approved therapy at least 4 weeks prior to Day 1 or drug-specific, 5 half-lives elimination period if longer than 4 weeks), and with no current plans to restart treatment during trial participation
   * Participants receiving any additional agent for IPF therapy must be on a stable regimen for at least 3 months prior to Day 1 with no current plans to change the treatment regimen during trial participation. Any previously discontinued therapy used to treat IPF must have been discontinued at least 4 weeks prior to Day 1 or 5 half-lives for that specific therapy must have elapsed, whichever is longer, with no plans to restart the therapy during trial participation.
4. Lung high-resolution computed tomography (HRCT) historically performed within 6 months prior to the Screening Visit and according to the minimum requirements for IPF diagnosis by central review based on participant's HRCT. If an evaluable HRCT is not available within 6 months prior to Screening, an HRCT will be performed at Screening to determine eligibility, according to the same requirements as the historical HRCT.
5. HRCT shows ≥10% to <50% parenchymal fibrosis (reticulation) and the extent of fibrotic changes is greater than the extent of emphysema on the most recent HRCT scan (central reviewer determined).
6. Meets all of the following criteria during the Screening Period:

   1. FVC ≥45% predicted of normal
   2. forced expiratory volume in 1 second (FEV1)/FVC ≥0.7
   3. Diffusing capacity of the lungs for carbon monoxide (DLCO) corrected for hemoglobin is ≥25% and ≤90% predicted of normal
7. Estimated minimum life expectancy of ≥30 months for non-IPF-related disease, in the opinion of the Investigator.
8. Vaccinations are up to date given age, comorbidities and local availability prior to trial drug dosing.
9. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the trial.

Key Inclusion Criteria in Extension Phase:

1. Completed the Double-blind Treatment Period (Week 52) of the Core Phase of the trial; subjects prematurely discontinued from trial drug in the Core Phase of the trial for reasons other than safety or tolerability may be included at the discretion of the Investigator after completing scheduled visits, including Week 52 assessments.
2. Willing and able to comply with the prescribed treatment protocol and evaluations for the duration of the Extension Phase of the trial.

Key Exclusion Criteria Core Phase:

1. Any of the following cardiovascular diseases:

   1. uncontrolled, severe hypertension (≥160/100 mmHg), within 6 months of Screening
   2. myocardial infarction within 6 months of Screening
   3. unstable cardiac angina within 6 months of Screening
2. Interstitial lung disease (ILD) associated with known primary diseases (e.g., sarcoidosis, amyloidosis and coronavirus disease 2019 [COVID-19]), connective tissue disorders (e.g., rheumatoid arthritis, systemic lupus erythematosus, Sjogren's, dermatomyositis, scleroderma), exposures (e.g., radiation, silica, asbestos and coal dust) or drugs (e.g., amiodarone).
3. Known active bacterial, viral, fungal, mycobacterial or other infection, including tuberculosis or atypical mycobacterial disease (fungal infections of nail beds are allowed). The participant must be 3 months beyond any acute infection with COVID-19 if there has been a prior infection.
4. Clinically significant pulmonary hypertension requiring chronic medical therapy.
5. Use of any of the following therapies within 4 weeks prior to Screening, during the Screening Period or planned during the trial: prednisone at steady dose >10 mg/day or equivalent or cyclosporine. Change in regimen or dosage of any immunosuppressant during the Screening Period through the end of trial participation will require consultation with and approval by the trial Medical Monitor.
6. Use of rifampin within 2 weeks prior to Day 1 or planned during the trial.
7. Malignant condition in the past 5 years (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
8. Women of childbearing potential (WOCBP) or male subjects not agreeing to use highly effective method(s) of birth control throughout the trial and for 4 weeks after last dose of trial drug. Females must refrain from egg/ova donation for 4 weeks after the last dose of trial drug and males must refrain from sperm donation for 3 months after the last dose of trial drug.
9. Pregnant or lactating women and women who plan to become pregnant or breast feed during the trial and within 4 weeks after the last dose of trial drug.
10. Current drug or alcohol abuse or history of either within the previous 2 years, in the opinion of the Investigator or as reported by the subject.
11. Previous enrollment in this trial or participation in a prior HZN-825 or SAR100842 clinical trial.
12. Known history of positive test for human immunodeficiency virus (HIV).
13. Active hepatitis (hepatitis B: positive hepatitis B surface antigen and positive anti-hepatitis B core antibody [anti-HBcAb] and negative hepatitis B surface antibody [HBsAb] or positive for HBcAb with a positive test for HBsAb and with presence of hepatitis B virus DNA at Screening; hepatitis C: positive anti-hepatitis C virus [anti-HCV] and positive RNA HCV).
14. Current alcoholic liver disease, primary biliary cirrhosis or primary sclerosing cholangitis.
15. Previous organ transplant (including allogeneic and autologous marrow transplant).
16. International normalized ratio >2, prolonged prothrombin time >1.5 × the upper limit of normal (ULN) or partial thromboplastin time >1.5 × ULN at Screening.
17. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.0 × ULN.
18. Estimated glomerular filtration rate <30 mL/min/1.73 m^2 at Screening.
19. Total bilirubin >1.5 × ULN. Subjects with documented diagnosis of Gilbert's syndrome may be enrolled if their total bilirubin is ≤3.0 mg/dL.
20. Moderate (Child-Pugh B) to severe (Child-Pugh C) hepatic impairment according to the Child-Pugh scoring system.
21. Any confirmed Grade 3 or higher laboratory abnormality.
22. Any laboratory abnormality at Screening that, in the opinion of the Investigator, would preclude the participant's entry in the trial.
23. Exposure to an experimental drug (with the exception of HZN-825) or experimental vaccine within either 30 days, 5 half-lives of the test agent, or twice the duration of the biological effect of the test agent, whichever is the longest, prior to Day 1.
24. Any other condition that, in the opinion of the Investigator, would preclude enrollment in the trial.

Key Exclusion Criteria Extension Phase:

1. Anticipated use of another investigational agent for any condition during the course of the trial.
2. New diagnosis of malignant condition after enrolling in Trial HZNP-HZN-825-303 (except successfully treated basal/squamous cell carcinoma of the skin or cervical cancer in situ).
3. Estimated minimum life expectancy ≤18 months, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (82):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Palmtree Clinical Research, Palm Springs, California
  - St. Francis Medical Institute, Clearwater, Florida
  - Central Florida Pulmonary Group PA, Orlando, Florida
  - DBC Research Corp., Tamarac, Florida
  - GCP Clinical Research, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Nebraska Pulmonary Specialties LLC, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Stony Brook Medicine Advanced Specialty Care, Commack, New York
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Shelby Clinical Research, Shelby, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - El Paso Pulmonary Association - Elligo, El Paso, Texas
  - Metroplex Pulmonary and Sleep Medicine Center, McKinney, Texas
  - Northwestern Memorial Hospital, Milwaukee, Wisconsin
- Argentina (6):
  - STAT Research S.A., Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Ave Pulmo, Mar del Plata, Buenos Aires
  - Instituto De Enfermedades Respiratorias E Investigacion Medica, San Juan Bautista, Buenos Aires
  - Instituto De Patologías Respiratorias, San Miguel de Tucumán, Tucumán Province
  - Centro Medico Dra de Salvo, Ciudad de Buenos Aires
  - Instituto Del Buen Aire, Santa Fe
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
- Canada (2):
  - Dynamic Drug Advancement Ltd., Ajax, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
- Chile (8):
  - Centro de Investigación Curico, Curicó, Maule Region
  - Centro Respiratorio Integral LTDA. (CENRESIN), Quillota, Región de Valparaíso
  - Universidad de Los Andes, Las Condes, Región-MetropolitanadeSantiago
  - MIRES/MYF estudios cli-nicos, Ñuñoa, Región-MetropolitanadeSantiago
  - Enroll SpA, Providencia, Región-MetropolitanadeSantiago
  - Meditek Ltda, Santiago, Región-MetropolitanadeSantiago
  - Centro de Investigacion del Maule, Talca
  - Clinical Research Chile SpA, Valdivia
- France (3):
  - Hopital Nord AP-HM, Marseille, Bouches-du-Rhône
  - Hopital Haut Leveque, Pessac, Gironde
  - Hôpital Bretonneau, Tours, Indre-et-Loire
- Lungenklinik Hemer, Hemer, North Rhine-Westphalia, Germany
- Greece (6):
  - University General Hospital of Patras, Pátrai, Achaïa
  - Evangelismos General Hospital of Athens, Athens, Attica
  - Athens Medical Center, Marousi, Attica
  - University General Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
- Italy (2):
  - Presidio Ospedaliero GB Morgagni L Pierantoni, Forlì, Emilia-Romagna
  - Azienda Ospedaliera Universitaria Senese, Siena
- Japan (6):
  - National Hospital Organization Himeji Medical Center, Himeji-Shi, Hyôgo
  - National Hospital Organization Ibarakihigashi National Hospital, Naka-Gun, Ibaraki
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Hiroshima Prefectural Hospital, Hiroshima
  - Medical Hospital of Tokyo Medical and Dental University, Tokyo
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakaishi, Ôsaka
- Mexico (4):
  - CICUM San Miguel, Guadalajara, Jalisco
  - Hospital Universitario Dr. Jose Eleuterio González, Monterrey, Nuevo León
  - Unidad de Investigación Clínica En Medicina SC, Monterrey, Nuevo León
  - Oaxaca Site management Organization (OSMO), Centro, Oaxaca
- Erasmus MC, Rotterdam, Netherlands
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - PULMAG Grzegorz Gasior Marzena Kociolek Spolka Cywilna, Katowice, Silesian Voivodeship
  - MCM Krakow - PRATIA - PPDS, Krakow
- South Africa (3):
  - KwaPhila Health Solutions, Durban, KwaZulu-Natal
  - University of Cape Town Lung Institute (UCTLI), Cape Town, Western Cape
  - Dr. Ismail Abdullah Private Practice, Cape Town, Western Cape
- South Korea (4):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Korea University Anam Hospital, Seoul
  - Asan Medical Center-PPDS, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (4):
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital - PPDS, Taichung
  - Far Eastern Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)
- Connolly Hospital Blanchardstown, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 153 participants with Idiopathic Pulmonary Fibrosis (IPF) were enrolled in 16 countries between January 2022 and December 2024.
Pre-assignment Details: This trial consisted of 2 parts. During part 1 (Core Phase) participants were randomized in 1:1:1 ratio to receive HZN-825 300 mg once daily (QD), twice daily (BID) or placebo, for 52 weeks. Part 2 (Extension Phase) was an optional, open-label extension (OLE) where all participants received HZN-825 BID for 52 weeks. 11 participants who completed part 1 did not enter the part 2.
Groups:
- HZN-825 300 mg QD Then HZN-825 300 mg BID: In the core phase participants received HZN-825 300 mg QD, for 52 weeks. In the optional OLE phase of the study (Part 2) participants received HZN-825 BID for 52 weeks.
- HZN-825 300 mg BID: In the core phase participants received HZN-825 300 mg BID, for 52 weeks. In the optional OLE phase of the study (Part 2) participants continued to receive HZN-825 BID for 52 weeks.
- Placebo Then HZN-825 300 mg BID: In the core phase participants received Placebo for 52 weeks. In the OLE phase of the study (Part 2) participants received HZN-825 BID for 52 weeks.
Period: Part 1: Core Phase
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Started | 49 | 52 | 52
Completed | 40 | 38 | 43
Not Completed | 9 | 14 | 9
Not completed — Withdrawal by Subject/Guardian | 4 | 6 | 5
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Death | 3 | 4 | 2
Not completed — Adverse Event | 2 | 3 | 0
Period: Part 2: Extension Phase
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Started | 36 | 34 | 40
Completed | 4 | 5 | 6
Not Completed | 32 | 29 | 34
Not completed — Withdrawal by Subject/Guardian | 2 | 1 | 2
Not completed — Study Terminated by Sponsor | 27 | 22 | 27
Not completed — Physician Decision | 1 | 2 | 0
Not completed — Death | 2 | 4 | 5

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who were randomized to a treatment and took at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID | Total
Number analyzed (Participants) | 49 | 52 | 52 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 7 | 31
  >=65 years | 35 | 42 | 45 | 122
Age, Continuous [Median (Full Range); unit: years] | 70.0 [50 to 82] | 73.5 [49 to 91] | 73.0 [58 to 81] | 73.0 [49 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 12 | 15 | 52
  Male | 24 | 40 | 37 | 101
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 16 | 25 | 67
  Not Hispanic or Latino | 23 | 36 | 27 | 86
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 12 | 16 | 9 | 37
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1
  White | 35 | 35 | 40 | 110
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1 | 2
Forced Vital Capacity (FVC) percent (FVC %) Predicted at Baseline [Mean (Standard Deviation); unit: % predicted FVC] — FVC was assessed using a blowing device provided by the Sponsor. The best of 3 efforts was defined as the highest FVC, obtained on any of the 3 blows meeting the American Thoracic Society (ATS)/European Respiratory Society (ERS) criteria with a maximum of 8 maneuvers.
  FVC % predicted was calculated by taking the observed FVC measurement and dividing it by a predicted value multiplied by 100 (% FVC predicted = (FVC observed/FVC predicted) x 100). The predicted value is an average of the normal FVC volume for a person of the same sex, ethnicity, age and height.
  % predicted FVC | 73.23 (17.074) | 72.11 (16.558) | 72.66 (12.761) | 72.66 (15.456)

OUTCOME MEASURES:

1. Primary Outcome: Core Phase: Change in FVC % Predicted From Baseline to Week 52
Description: FVC was assessed using a blowing device provided by the Sponsor. The best of 3 efforts was defined as the highest FVC, obtained on any of the 3 blows meeting the ATS/ERS criteria with a maximum of 8 maneuvers.
  FVC % predicted was calculated by taking the observed FVC measurement and dividing it by a predicted value multiplied by 100 (% FVC predicted = (FVC observed/FVC predicted) x 100). The predicted value is an average of the normal FVC volume for a person of the same sex, ethnicity, age and height.
Time Frame: Baseline and Week 52
Population: Full Analysis Set (FAS): All participants who were randomized and took at least 1 dose of HZN-825.
Measure: Least Squares Mean (Standard Error); unit: % predicted FVC
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
% predicted FVC | -4.13 (1.045) | -3.38 (1.092) | -2.99 (1.025)
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; The primary analysis was based on a mixed model for repeated measures (MMRM) analysis of covariance (ANCOVA) model using observed change in FVC % predicted values from all planned post-baseline assessments (Weeks 4, 16, 28, 40 and 52) with covariates of treatment group (300 mg HZN-825 QD, 300 mg HZN-825 BID, placebo), prior use of IPF therapy [yes or no], FVC% predicted at baseline [≥ 70, <70], visit week, and treatment by visit week interaction; Test type: Superiority; p = 0.4388, Mixed Model for Repeated Measures (MMRM); Least Squares (LS) Mean Difference = -1.13, 90% CI 2-sided [-3.56 to 1.29], Standard Error of Mean 1.460
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7959, MMRM; LS Mean Difference = -0.39, 90% CI 2-sided [-2.86 to 2.09], Standard Error of Mean 1.493

2. Primary Outcome: Extension Phase: Change in FVC % Predicted From OLE Baseline to Week 104
Description: OLE baseline was defined as the latest measurement prior to the first dose of HZN-825 in the extension phase.
  FVC was assessed using a blowing device provided by the Sponsor. The best of 3 efforts was defined as the highest FVC, obtained on any of the 3 blows meeting the ATS/ERS criteria with a maximum of 8 maneuvers.
  FVC % predicted was calculated by taking the observed FVC measurement and dividing it by a predicted value multiplied by 100 (% FVC predicted = (FVC observed/FVC predicted) x 100). The predicted value is an average of the normal FVC volume for a person of the same sex, ethnicity, age and height.
Time Frame: OLE baseline (Week 52) and Week 104
Population: OLE Phase Analysis Set (OLE-SAF): All participants that were enrolled in OLE Phase and took at least 1 dose of HZN-825 during the OLE Phase.
Measure: Mean (Standard Deviation); unit: % predicted FVC
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 4 | 3 | 5
% predicted FVC | 11.38 (23.237) | -0.63 (16.283) | -2.62 (6.305)

3. Secondary Outcome: Core Phase: Number of Participants With a Decline in FVC % Predicted ≥10% From Baseline at Week 52
Description: as for outcome 1
Time Frame: Baseline and Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825.
Measure: Number; unit: participants
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
participants | 6 | 7 | 4
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; The percentage of participants with a decrease in FVC% predicted ≥10% from baseline at Week 52 were analyzed with observed data using a stratified logistic regression model. Baseline value and treatment were considered as factors in the model and prior use of approved IPF therapy [yes or no], FVC% predicted at baseline [≥ 70, <70] were considered as stratification factors; Test type: Superiority; p = 0.7179, Stratified logistic regression; Odds Ratio (OR) = 0.854, 90% CI 2-sided [0.417 to 1.750]
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0706, Stratified logistic regression; Odds Ratio (OR) = 0.469, 90% CI 2-sided [0.236 to 0.934]

4. Secondary Outcome: Core Phase: Change in the 6-Minute Walk Test (6MWT) Results From Baseline to Week 52
Description: The 6MWT measures the distance a subject can quickly walk on a flat, hard surface in 6 minutes (6-minute walk distance). This test evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units and muscle metabolism.
Time Frame: Baseline and Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Meters | 14.00 (12.990) | -3.95 (13.081) | -2.71 (12.757)
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; Estimated from a mixed effect repeated measurement analysis with unstructured variance-covariance matrix, that included factors treatment (300 mg HZN-825 QD, 300 mg HZN-825 BID, placebo), the Baseline factors used for stratifying randomization as covariates (prior use of approved IPF therapy [yes/no] and Baseline FVC% Predicted [>=70, <70], as used in IRT randomization), visit week, and treatment by visit week interaction; Test type: Superiority; p = 0.3579, MMRM; LS Mean Difference = 16.71, 90% CI 2-sided [-13.30 to 46.73], Standard Error of Mean 18.109
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.9460, MMRM; LS Mean Difference = -1.23, 90% CI 2-sided [-31.35 to 28.88], Standard Error of Mean 18.173

5. Secondary Outcome: Core Phase: Change in King's Brief Interstitial Lung Disease (K-BILD) Questionnaire Scores From Baseline to Week 52
Description: The K-BILD is a self-completed health status questionnaire comprising 15 items and a 7-point Likert response scale that was developed and validated specifically for patients with IPF. This questionnaire has 3 domains: psychological, breathlessness and activities and chest symptoms. The K-BILD domains and total score range from 0 to 100; 100 represents best health status. A positive change from baseline indicates an improvement in symptoms.
Time Frame: Baseline and Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Score on a scale | -1.5 (1.65) | -1.4 (1.67) | -0.3 (1.62)
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; Estimated from a MMRM with unstructured variance-covariance matrix, that included treatment group, time point, treatment by timepoint interaction, and stratification factors as covariates; Test type: Superiority; p = 0.6091, MMRM; LS Mean Difference = -1.2, 90% CI 2-sided [-5.0 to 2.6], Standard Error of Mean 2.30
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.6374, MMRM; LS Mean Difference = -1.1, 90% CI 2-sided [-4.9 to 2.7], Standard Error of Mean 2.31

6. Secondary Outcome: Core Phase: Change in Living With IPF (L-IPF) Scores From Baseline to Week 52
Description: The L-IPF is a validated questionnaire that assesses symptoms, disease impacts and health-related quality of life in subjects with IPF. This questionnaire was developed with input from the FDA and comprises 2 modules: a 15-item symptom module with 3 domains (dyspnea, cough, and energy), all with a 24-hour recall, and a 20-item impacts module with 1-week recall. Symptoms Total Score and Impacts Total Score were transformed to a model-based scale ranging from 0 to 100 where higher scores indicate greater impairment.
Time Frame: Baseline and Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Score on a scale
  L-IPF Symptoms Total Score | 4.0 (1.42) | 2.6 (1.45) | 0.6 (1.39)
  L-IPF Impact Total Score | 3.1 (1.93) | 1.3 (1.97) | -0.8 (1.90)
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; Impact Total Score Estimated from a mixed effect repeated measurement analysis with unstructured variance-covariance matrix, that included factors baseline FVC% predicted, treatment (300 mg HZN-825 QD, 300 mg HZN-825 BID, placebo), the Baseline factors used for stratifying randomization as covariates (prior use of approved IPF therapy [yes/no] and Baseline FVC% Predicted [>=70, <70]), visit week, and treatment by visit week interaction; Test type: Superiority; p = 0.1526, MMRM; LS Mean Difference = 3.9, 90% CI 2-sided [-0.6 to 8.3], Standard Error of Mean 2.69
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.4421, MMRM; LS Mean Difference = 2.1, 90% CI 2-sided [-2.4 to 6.6], Standard Error of Mean 2.72
Statistical Analysis 3: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; Symptoms Total Score Estimated from a mixed effect repeated measurement analysis with unstructured variance-covariance matrix, that included factors baseline FVC% predicted, treatment (300 mg HZN-825 QD, 300 mg HZN-825 BID, placebo), the Baseline factors used for stratifying randomization as covariates (prior use of approved IPF therapy [yes/no] and Baseline FVC% Predicted [>=70, <70]), visit week, and treatment by visit week interaction; Test type: Superiority; p = 0.0936, MMRM; LS Mean Difference = 3.3, 90% CI 2-sided [0.1 to 6.6], Standard Error of Mean 1.98
Statistical Analysis 4: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 6, analysis 3]; Test type: Superiority; p = 0.3129, MMRM; LS Mean Difference = 2.0, 90% CI 2-sided [-1.3 to 5.3], Standard Error of Mean 2.00

7. Secondary Outcome: Core Phase: Change in Leicester Cough Questionnaire (LCQ) Scores From Baseline to Week 52
Description: The LCQ is a patient-reported questionnaire evaluating the impact of cough on quality of life. The LCQ comprises 19 items and takes 5 to 10 minutes to complete. Each item assesses symptoms or the impact of symptoms over the last 2 weeks on a 7-point Likert scale. Scores in 3 domains (physical, psychological, and social) are calculated as a mean for each domain (range: 1 to 7). A total score (range: 3 to 21) is also calculated by adding together the domain scores. Higher scores indicate better quality of life and a positive change from baseline indicates an improvement in quality of life.
Time Frame: Baseline to Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Score on a scale | 0.19 (0.463) | -0.45 (0.468) | 0.54 (0.453)
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; Estimated from a mixed effect repeated measurement analysis with unstructured variance-covariance matrix, that included factors baseline FVC% predicted, treatment (300 mg HZN-825 QD, 300 mg HZN-825 BID, placebo), the Baseline factors used for stratifying randomization as covariates (prior use of approved IPF therapy [yes/no] and Baseline FVC% Predicted [>=70, <70]), visit week, and treatment by visit week interaction; Test type: Superiority; p = 0.5832, MMRM; LS Mean Difference = -0.35, 90% CI 2-sided [-1.42 to 0.71], Standard Error of Mean 0.644
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 7, analysis 1]; Test type: Superiority; p = 0.1297, MMRM; LS Mean Difference = -0.99, 90% CI 2-sided [-2.06 to 0.09], Standard Error of Mean 0.648

8. Secondary Outcome: Core Phase: Time to First Hospitalization Due to Respiratory Distress From Baseline up to Week 52
Description: Hospitalization due to respiratory distress was defined as a non-elective hospitalization lasting more than 24 hours in a hospital, emergency room or observation unit, due to respiratory causes that occur after randomization Adverse events identified as leading to hospitalization due to respiratory distress were adjudicated to confirm that the event and hospitalization met the stated criteria. Participants who did not experience a hospitilization event were considered censored.
Time Frame: Up to Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825, inclusive of censoring.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Days | NA [NA to NA] — Time to event was analyzed using the Kaplan-Meier method, but the median and inter-quartile range (IQR) could not be estimated due to limited number of events at the time of analysis. | NA [NA to NA] — Time to event was analyzed using the Kaplan-Meier method, but the median and IQR could not be estimated due to limited number of events at the time of analysis. | NA [NA to NA] — Time to event was analyzed using the Kaplan-Meier method, but the median and IQR could not be estimated due to limited number of events at the time of analysis.
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; Estimated from a stratified Cox proportional hazards regression model stratified by prior use of approved IPF therapy [yes or no] and FVC% predicted at baseline [= 70, <70] and treatment group as factor. Placebo group is the reference group for the analysis; Test type: Superiority; p = 0.9996, Regression, Cox; Hazard Ratio (HR) = 1.00, 90% CI 2-sided [0.34 to 2.90]
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3721, Regression, Cox; Hazard Ratio (HR) = 1.66, 90% CI 2-sided [0.66 to 4.48]

9. Secondary Outcome: Core Phase: Time to First Onset of the Composite Endpoint of Progression-Free Survival (PFS) From Baseline up to Week 52
Description: The time-to-progression was defined as the duration from the date of first dose of study drug to either (a) the date of the visit where FVC % predicted declines ≥ 10% from Baseline or (b) the date of participant death, whichever occurred earlier. Results were given based on the Kaplan-Meier reading with a cutoff at Day 365.
Time Frame: Up to Week 52
Population: FAS: All participants who were randomized and took at least 1 dose of HZN-825, inclusive of censoring.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Days | NA [NA to NA] — There was an insufficient number of participants with an event to calculate the upper limit. The results for the median and lower limit were beyond the cutoff date of Day 365. | NA [357 to NA] — The results for the median and upper limit were beyond the cutoff date of Day 365. | NA [NA to NA] — There was an insufficient number of participants with an event (7) to calculate a median and inter-quartile range.
Statistical Analysis 1: Comparison: HZN-825 300 mg QD Then HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.4778, Regression, Cox; Hazard Ratio (HR) = 1.42, 90% CI 2-sided [0.63 to 3.32]
Statistical Analysis 2: Comparison: HZN-825 300 mg BID vs Placebo Then HZN-825 300 mg BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0438, Regression, Cox; Hazard Ratio (HR) = 2.52, 90% CI 2-sided [1.22 to 5.61]

10. Secondary Outcome: Core Phase: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A TEAE was considered a serious adverse event (SAE) if it resulted in any of the following: death; life-threatening experience; persistent or significant disability or incapacity; inpatient hospitalization or prolongation of hospitalization; congenital anomaly or birth defect; medically important event that may require medical or surgical intervention to prevent one of the outcomes listed. An adverse event of special interest (AESI) was an AE of scientific and medical concern specific to HZN-825. Orthostatic hypotension was considered an AESI. Clinically significant changes in vital signs, electrocardiograms, echocardiograms and laboratory tests recorded after treatment administration were documented as TEAEs.
Time Frame: From 1st dose to last dose + 28 days, Median (min, max) duration was 12.0 (1.0, 13.1) months for Core Phase and 7.0 (1.6, 13.2) months for OLE Phase.
Population: Safety analysis set: all participants who took any dose of study drug during the Core Phase.
Measure: Number; unit: Participants
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID | Placebo Then HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52 | 52
Participants
  Core Phase: TEAEs | 38 | 42 | 38
  Core Phase: SAEs | 10 | 14 | 9
  Core Phase: AESIs | 1 | 2 | 1
  Extension Phase: TEAEs: number analyzed (Participants) | 36 | 34 | 40
  Extension Phase: TEAEs | 27 | 22 | 33
  Extension Phase: SAEs: number analyzed (Participants) | 36 | 34 | 40
  Extension Phase: SAEs | 8 | 6 | 9
  Extension Phase: AESIs: number analyzed (Participants) | 36 | 34 | 40
  Extension Phase: AESIs | 0 | 1 | 0

11. Secondary Outcome: Core Phase: Pre- and Post-dose Concentrations of HZN-825
Description: Pre- and Post-dose Concentrations of HZN-825 were presented.
Time Frame: Day 1 (2-4 hours after the first dose), Week 4 (pre-dose), Week 10, Weeks 16 and 28 (pre-dose and 2-4 hours post-dose), and Weeks 40 and 52 (pre-dose for participants entering OLE).
Population: Pharmacokinetic analysis set: all randomized participants who took at least 1 dose of HZN-825 and have at least 1 nonmissing postdose concentration value reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HZN-825 300 mg QD Then HZN-825 300 mg BID | HZN-825 300 mg BID
Number analyzed (Participants) | 49 | 52
ng/mL
  Day 1 (Post-dose): number analyzed (Participants) | 49 | 51
  Day 1 (Post-dose) | 16676.2 (11030.30) | 16209.4 (11592.69)
  Week 4 (Pre-dose): number analyzed (Participants) | 47 | 47
  Week 4 (Pre-dose) | 6521.3 (7756.18) | 18360.0 (11953.98)
  Week 10: number analyzed (Participants) | 45 | 46
  Week 10 | 11372.8 (11123.02) | 23807.8 (13864.61)
  Week 16 (Pre-dose): number analyzed (Participants) | 45 | 46
  Week 16 (Pre-dose) | 5296.4 (3093.68) | 16889.8 (9952.20)
  Week 16 (Post-dose): number analyzed (Participants) | 45 | 44
  Week 16 (Post-dose) | 21162.9 (11543.77) | 24629.3 (11871.17)
  Week 28 (Pre-dose): number analyzed (Participants) | 45 | 43
  Week 28 (Pre-dose) | 5435.8 (4125.22) | 19258.1 (10368.10)
  Week 28 (Post-dose): number analyzed (Participants) | 43 | 40
  Week 28 (Post-dose) | 19410.7 (13812.87) | 27598.4 (13634.06)
  Week 40 (Pre-dose): number analyzed (Participants) | 40 | 39
  Week 40 (Pre-dose) | 8487.6 (9209.61) | 20702.0 (13362.76)
  Week 52 (Pre-dose): number analyzed (Participants) | 42 | 38
  Week 52 (Pre-dose) | 5030.2 (3998.99) | 17330.1 (10638.75)

ADVERSE EVENTS:
Time Frame: Death: From randomization to end of study (EOS), Median (min, max) was 17.7 (0.1, 25.9) months. TEAE: From 1st dose to last dose + 28 days, Median (min, max) duration was 12.0 (1.0, 13.1) months for Core Phase and 7.0 (1.6, 13.2) months for OLE Phase.
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Core Phase: HZN-825 300mg QD: Participants received HZN-825 QD orally as two 150 mg tablets in the core phase.
- Core Phase: HZN-825 300mg BID: Participants received HZN-825 BID orally as two 150 mg tablets in the core phase.
- Core Phase: Placebo: Participants received matching placebo orally as tablets in the core phase.
- OLE Phase: HZN-825 300mg BID: All participants who received HZN-825 BID orally as two 150 mg tablets in the OLE Phase.
Arm/Group | Core Phase: HZN-825 300mg QD | Core Phase: HZN-825 300mg BID | Core Phase: Placebo | OLE Phase: HZN-825 300mg BID
All-Cause Mortality (participants affected / at risk) | 3/49 | 4/52 | 2/52 | 11/110
Serious Adverse Events (participants affected / at risk) | 10/49 | 14/52 | 9/52 | 23/110
Other Adverse Events (participants affected / at risk) | 23/49 | 33/52 | 20/52 | 35/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core Phase: HZN-825 300mg QD (N=49) | Core Phase: HZN-825 300mg BID (N=52) | Core Phase: Placebo (N=52) | OLE Phase: HZN-825 300mg BID (N=110)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Retinal artery thrombosis (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Gallbladder rupture (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic necrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 4
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 2 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Obstructive nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 5
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core Phase: HZN-825 300mg QD (N=49) | Core Phase: HZN-825 300mg BID (N=52) | Core Phase: Placebo (N=52) | OLE Phase: HZN-825 300mg BID (N=110)
Diarrhoea (Gastrointestinal disorders) | 5 | 1 | 5 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 3 | 2 | 7
Nasopharyngitis (Infections and infestations) | 4 | 3 | 4 | 7
Pneumonia (Infections and infestations) | 1 | 4 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 1 | 2
Urinary tract infection (Infections and infestations) | 6 | 3 | 2 | 7
Activated partial thromboplastin time prolonged (Investigations) | 1 | 4 | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 3
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 3
Headache (Nervous system disorders) | 1 | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2 | 2
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 1

LIMITATIONS AND CAVEATS:
The trial was terminated due to not meeting primary or key secondary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT05032066/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/66/NCT05032066/SAP_002.pdf